CLINICAL TRIAL: NCT02015611
Title: Trial of Vitamin D Supplementation and Neuromuscular Function in Older Adults
Brief Title: Vitamin D Supplementation and Muscle Function in Older Adults
Acronym: EVIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00022395; R01AG042411 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-09

CONDITIONS: Neuromuscular Function
Keywords: Vitamin D; Muscle power; Muscle fiber; Falls; Aging
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matched bottle/pill placebo
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Experimental): 2,000 IU Vitamin D3 per day
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 2,000 IU/ day of Vitamin D3
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if vitamin D supplementation improves muscle function in older adults.

DETAILED DESCRIPTION:
This study is a 12-month, double-blind randomized placebo controlled trial in older (65-89 yrs) men and women with initial 25(OH)D concentrations of 18-<30 ng/mL to determine the effect of increasing 25(OH)D concentrations to ≥30 ng/mL through vitamin D3 supplementation on 1) change in neuromuscular functions that are established risk-factors for falls in older adults; and 2) changes in the underlying physiological mechanisms over 4 months in a subset of randomly selected participants. Participants will be randomized to 2000 IU/d of vitamin D3 or placebo. Lower extremity muscle strength and power, physical performance, and postural sway will be assessed at baseline, 4 months and 12 months and falls assessed monthly. Muscle biopsies of the vastus lateralis will be taken at baseline and 4 months to assess muscle fiber type, contractility, and denervation, and number and differentiation stage of satellite cells.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 to <90 years
* SPPB <=10
* Initial serum 25(OH)D concentration of 18 to <30 ng/mL
* Not dependent on a walker
* Able to provide own transportation to study visits
* Not involved in another intervention study
* Willing to provide informed consent and adhere to the protocol

Exclusion Criteria:

* Serious or uncontrolled chronic disease including: insulin-dependent diabetes; cancer requiring treatment in past year, except non-melanoma skin cancers; acute coronary event (within the last 6 months), uncontrolled angina, heart failure (stage 3-4), PAD, or stroke (within the last 6 months); uncontrolled hypertension (BP>200/110 mmHg); chronic respiratory disease requiring the use of oxygen; uncontrolled endocrine/metabolic disease; neurological (e.g., Parkinson's disease) or hematological disease; liver or renal dysfunction (eGFR <45 mL/min/1.73m2); and musculoskeletal impairments severe enough to preclude functional testing
* Evidence of impaired cognitive function (MoCA <18)
* Taking prescription vitamin D2 or taking >1000 IU/day of vitamin D3 (from all sources); taking an oral corticosteroid (i.e., prednisone at 7.5mg/d for 3 mos or equivalent); taking hormone replacement therapy
* Inability or contraindications to consume daily vitamin D supplements (e.g., hypercalcemia, sarcoidosis, history of kidney stones in last 5 years)
* Knee or hip surgery within the last 6 months or planned knee or hip surgery within the next year
* Unwillingness to undergo a muscle biopsy or use of anti-coagulants
* Unintentional weight loss of ≥5% or more in the past 3 months
* BMI >40 kg/m2
* If the PI feels the participant is unlikely to follow the protocol

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise K Houston, PhD, RD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Houston DK, Marsh AP, Neiberg RH, Demons JL, Campos CL, Kritchevsky SB, Delbono O, Tooze JA. Vitamin D Supplementation and Muscle Power, Strength and Physical Performance in Older Adults: A Randomized Controlled Trial. Am J Clin Nutr. 2023 Jun;117(6):1086-1095. doi: 10.1016/j.ajcnut.2023.04.021. Epub 2023 Apr 19. PMID 37084814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 70 | 66
Completed | 65 | 64
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 70 | 66 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (6.3) | 73.7 (6.3) | 73.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 35 | 34 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 21 | 44
  White | 47 | 45 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Short Physical Performance Battery Score [Least Squares Mean (Standard Deviation); unit: score on a scale] — The scores range from 0 (worst performance) to 12 (best performance).
  score on a scale | 7.7 (0.2) | 7.7 (0.2) | 7.7 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Muscle Power Over 12 Months
Description: Lower extremity muscle power will be measured at baseline, 4- and 12-month follow-up using the Nottingham Power Rig. Participants sit in a chair and unilaterally depress a foot lever attached to a flywheel as hard and as fast as they can. Power output, derived from the acceleration of the flywheel from 5 trials on each leg at maximal effort, will be recorded in Watts. Maximum leg power at baseline (from either the right or left leg) and the maximum power from the same leg at 4- and 12-month follow-up will be used in all analyses. Leg power (Watts) will be standardized to total body mass (in Kg).
Time Frame: change from baseline at 12 month follow-up reported
Population: 4 participants in the placebo arm and 3 participants in the vitamin D arm were missing the leg power outcome at 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Watts/kg
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 61 | 61
Watts/kg | -0.10 (0.04) | -0.13 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.63, ANCOVA; adjusted for age, sex, race, season (time-varying)

2. Primary Outcome: Change in Percentage of Type II (Fast-twitch) Muscle Fibers Over 4 Months
Description: This will be examined in muscle biopsies collected at baseline and 4-month follow-up using the ATPase, pH 9.4 technique, combined with laminin immunostaining in 10 micrometer muscle sections and the number of type I and type II fiber subtypes quantified. The percentage of type II fibers is calculated by dividing the number of type II fibers by the sum of type I and type II fibers combined.
Time Frame: over 4 months of follow-up
Population: Subset of participants from main trial with muscle biopsy at baseline and 4 months
Measure: Least Squares Mean (Standard Error); unit: Percent of type II muscle fibers
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 14 | 18
Percent of type II muscle fibers | -1.35 (3.56) | -3.68 (2.81)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.64, Regression, Linear; adjusted for age, sex, race, season, and baseline value

3. Secondary Outcome: Change in Lower Extremity Muscle Strength Over 12 Months
Description: Lower extremity muscle strength will be measured using an isokinetic dynamometer (Biodex) at one speed (60°/sec) with the participant sitting and the hips and knee flexed at 90°. Participants extend the knee and push as hard as possible against the resistance pad. Strength is expressed as peak torque in Newton-meters (Nm). The maximum knee extensor strength of the 4 repetitions from trial 2 for the dominant leg will be will be used in analyses unless unable to test the dominant leg (i.e., knee replacement) in which case the non-dominant leg will be used; the maximum knee extensor strength from the same leg will be used at 4- and 12-month follow-up for all analyses.
Time Frame: change from baseline at 12 month follow-up reported
Population: Participants excluded from testing if they had ever had knee surgery, had difficulty bending/straightening either of their knees fully due to pain, arthritis, injury, or other condition, or experienced pain upon testing. At baseline, only 60 participants in the placebo group and 55 participants in the vitamin D group were able to test. At 12-month follow-up, only 50 participants in the placebo and 45 participants in the vitamin D group were able to test.
Measure: Least Squares Mean (Standard Error); unit: Newton meters
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 50 | 45
Newton meters | -3.84 (1.66) | -8.09 (1.75)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.08, ANCOVA; adjusted for age, sex, race, season (time-varying)

4. Secondary Outcome: Change in the Short Physical Performance Battery (SPPB) Score Over 12 Months
Description: The short physical performance battery consists of standing balance (side-by-side, semi- and full-tandem stands for 10 seconds), a 4-m walk to assess usual gait speed, and 5 repeated chair stands at baseline, 4-months and 12-months. Each of the three performance measures is assigned a score ranging from 0 (inability to perform the task) to 4 (the highest level of performance) and summed to create an SPPB score ranging from 0 to 12 (best).
Time Frame: change from baseline at 12 month follow-up reported
Population: 2 participants in the placebo group and 4 in the vitamin D group were excluded from analyses: 4 participants because they used an assistive device during testing at follow-up but not at baseline (1 in the placebo group and 3 in the vitamin D group); 1 participant because of severe knee pain and limping at follow-up (placebo group); and 1 participant was in a walking boot at 12-month follow-up (vitamin D group).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 63 | 60
score on a scale | 1.83 (0.22) | 1.64 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.53, ANCOVA; adjusted for age, sex, race, season (time-varying)

5. Secondary Outcome: Change in the Expanded Physical Performance Battery Score Over 12 Months
Description: The expanded physical performance battery consists of standing balance (semi- and full-tandem stands and a single leg stand for 30 seconds), a 4-m walk to assess usual gait speed, a narrow 4-m walk test of balance (walking at usual pace within lines of tape spaced 20 cm apart), and 5 repeated chair stands at baseline, 4-months, and 12-months. Scores range from 0 to 4 with higher scores indicative of better physical performance.
Time Frame: change from baseline at 12 month follow-up reported
Population: 14 participants in the placebo group and 10 in the vitamin D group were excluded from analyses: 4 participants because they used an assistive device during testing at follow-up but not at baseline (1 in the placebo group and 3 in the vitamin D group); 1 participant because of severe knee pain and limping at follow-up (placebo group); 1 participant was in a walking boot at 12-month follow-up (vitamin D group); and 12 in the placebo group and 6 in the vitamin D group due to change >2 IQR
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 51 | 54
score on a scale | 0.17 (0.04) | 0.19 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.75, ANCOVA; adjusted for age, sex, race, season (time-varying)

6. Secondary Outcome: Change in Timed Up and Go (TUG) Over 12 Months
Description: The timed up and go will be measured by how long it takes (sec) to stand up from a chair, walk 3 m, turn around, walk back to the chair, and sit down at baseline, 4-months, and 12-months. Longer times to complete the TUG are indicative of greater fall risk.
Time Frame: change from baseline at 12 month follow-up reported
Population: 6 participants in the placebo group and 6 in the vitamin D group were excluded from analyses due to: 1 participant with foot pain (placebo group), 1 participant with knee pain and limping (placebo group), 3 participants using an aid at follow-up but not at baseline (2 placebo and 1 vitamin D group), 1 participant with vertigo (placebo group), and 6 participants with change >2 IQR (1 placebo group, 5 vitamin D group)
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 59 | 58
seconds | 0.98 (0.21) | 1.01 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.92, ANCOVA; adjusted for age, sex, race, season (time-varying)

7. Secondary Outcome: Change in Average Sway Velocity Over 12 Months
Description: Postural sway during quiet stance will be assessed from Center-of-Pressure (COP) trajectory data collected at 100 Hz using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform at baseline, 4-months, and 12-months. Participants stand on the force platform barefoot in an upright stance with arms relaxed comfortably at their sides, eyes open, feet abducted 10 degrees, and heels separated medio-laterally by 6 cm. COP data is collected in a series of 10 30-sec trials standing on the force plate. Average sway velocity is measured in cm/sec. A higher number indicates more postural sway.
Time Frame: change from baseline at 12 month follow-up reported
Population: 14 participants in the placebo group and 10 in the vitamin D group were excluded from analysis: 1 participant with a foot in a walking boot (vitamin D group), 1 participant with foot pain (placebo group), 1 participant with severe knee pain (placebo group), and 12 in the placebo group and 9 in the vitamin D group due to change >2 IQR
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 51 | 54
cm/sec | 0.01 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.94, ANCOVA; adjusted for age, sex, race, season (time-varying)

8. Secondary Outcome: Change in 95% Confidence Ellipse Area Over 12 Months
Description: Postural sway during quiet stance will be assessed from Center-of-Pressure (COP) trajectory data collected at 100 Hz using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform at baseline, 4-months, and 12-month. Participants stand on the force platform barefoot in an upright stance with arms relaxed comfortably at their sides, eyes open, feet abducted 10 degrees, and heels separated medio-laterally by 6 cm. COP data is collected in a series of 10 30-sec trials standing on the force plate. 95% confidence ellipse area is measured in cm squared. A higher number indicates more postural sway.
Time Frame: change from baseline at 12 month follow-up reported
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: cm squared
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 51 | 54
cm squared | 0.00 (0.04) | 0.03 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.61, ANCOVA; adjusted for age, sex, race, season (time-varying)

9. Secondary Outcome: Change in Maximum Anteroposterior (AP) Displacement Over 12 Months
Description: Postural sway during quiet stance will be assessed from Center-of-Pressure (COP) trajectory data collected at 100 Hz using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform at baseline, 4-months, and 12-months. Participants stand on the force platform barefoot in an upright stance with arms relaxed comfortably at their sides, eyes open, feet abducted 10 degrees, and heels separated medio-laterally by 6 cm. COP data is collected in a series of 10 30-sec trials standing on the force plate. Anteroposterior (AP) displacement is measured in cm. A higher number indicates more postural sway.
Time Frame: change from baseline at 12 month follow-up reported
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 51 | 54
cm | 0.00 (0.03) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.59, ANCOVA; adjusted for age, sex, race, season (time-varying)

10. Secondary Outcome: Change in Maximum Mediolateral (ML) Displacement Over 12 Months
Description: Postural sway during quiet stance will be assessed from Center-of-Pressure (COP) trajectory data collected at 100 Hz using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform at baseline, 4-months, and 12-months. Participants stand on the force platform barefoot in an upright stance with arms relaxed comfortably at their sides, eyes open, feet abducted 10 degrees, and heels separated medio-laterally by 6 cm. COP data is collected in a series of 10 30-sec trials standing on the force plate. Mediolateral (ML) displacement is measured in cm. A higher number indicates more postural sway.
Time Frame: change from baseline at 12 month follow-up reported
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 51 | 54
cm | -0.01 (0.04) | 0.06 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority; p = 0.21, ANCOVA; adjusted for age, sex, race, season (time-varying)

11. Other Pre Specified Outcome: Number of Falls Over 12 Months
Description: Falls will be defined as an event whereby an individual unexpectedly comes to rest on the ground or another lower level. Participants will be provided monthly fall calendars and asked to mark any falls that occur on the calendar. Completion of monthly fall calendars will be monitored via monthly phone calls and collected at the 4- and 12-month visits. The number of total falls per participant over the entire 12-month follow-up period will be used in analysis.
Time Frame: monthly over 12 months
Population: 1 participant in the placebo group and 4 participants in the vitamin D group did not return their falls calendar
Measure: Mean (Standard Deviation); unit: number of falls
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 64 | 60
number of falls | 1.47 (2.76) | 1.40 (2.85)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/66
Serious Adverse Events (participants affected / at risk) | 12/70 | 6/66
Other Adverse Events (participants affected / at risk) | 29/70 | 16/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | Vitamin D (N=66)
Hospitalization (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization (Cardiac disorders) | 2 (2) | 1 (1)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalization (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hospitalization (Immune system disorders) | 1 (1) | 0 (0)
Hospitalization (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hospitalization (Infections and infestations) | 3 (4) | 2 (3)
Life threatening illness or accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization (Renal and urinary disorders) | 1 (3) | 0 (0)
Hospitalization (Surgical and medical procedures) | 2 (2) | 1 (3)
Hospitalization (Vascular disorders) | 0 (0) | 1 (1)
Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | Vitamin D (N=66)
Arthritis (Musculoskeletal and connective tissue disorders) | 10 (10) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 8 (10) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT02015611/Prot_SAP_000.pdf